CLINICAL TRIAL: NCT02597582
Title: A Prospective Randomized Study of LigaSure Small Jaw® Versus Conventional Neck Dissection in Head and Neck Cancer Patients
Brief Title: LigaSure Small Jaw® Versus Conventional Neck Dissection in Head and Neck Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Shih-An Liu, Attending physician, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: TCVGH-1037004C
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Head and Neck Neoplasms
Keywords: LigaSure; Neck dissection; Operative duration; Postoperative drainage; Postoperative pain
MeSH Terms: conditions — Head and Neck Neoplasms; Pain, Postoperative | interventions — Neck Dissection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ligusure assisted neck dissection (Active Comparator): The study group patients were treated using the LigaSure vessel sealing system (Small Jaw® with ForceTriad®; Covidien, Colorado, USA) for dissection and hemostasis throughout the whole procedures during neck dissection.
  Participants were asked to take a Voren enteric-microencapsulated (Diclofenac 50 mg/capsule) capsule 3 times a day for pain relief postoperatively. An additional capsule before sleep was allowed if persistent pain was told by the patient. When intolerable pain was complained in spite of oral analgesic, pethidine (meperidine 50 mg/ampule) injection was prescribed every 6 hours.
  Interventions: Procedure: Neck dissection
- Conventional neck dissection (Other): The control group patients were treated using conventional cold instrument dissection, monopolar electrocautery hemostasis, and suture ligation during neck dissection.
  Participants were asked to take a Voren enteric-microencapsulated (Diclofenac 50 mg/capsule) capsule 3 times a day for pain relief postoperatively. An additional capsule before sleep was allowed if persistent pain was told by the patient. When intolerable pain was complained in spite of oral analgesic, pethidine (meperidine 50 mg/ampule) injection was prescribed every 6 hours.
  Interventions: Procedure: Neck dissection

INTERVENTIONS:
Procedure: Neck dissection — The Small Jaw® handpiece (Small Jaw® with ForceTriad®; Covidien, Colorado, USA) was not only used as a dissection forceps but also served as a ligation device.
  Other Names: Ligasure vessel sealing system

SUMMARY:
The aim of this prospective randomized study was to investigate if the LigaSure vessel sealing system can reduce the operation duration and the postoperative drainage amount in patients undergoing neck dissection.

DETAILED DESCRIPTION:
We compared the differences in perioperative and postoperative variables between LigaSure Small Jaw®-assisted and conventional neck dissection in head and neck cancer patients.

Patients who were scheduled to undergo neck dissection due to head and neck cancer were eligible for this study. After receiving a detailed explanation, all patients signed an informed consent form before randomization. The study group were treated using the LigaSure vessel sealing system (Small Jaw®; Covidien, Colorado, USA) for dissection and hemostasis throughout the whole procedures during neck dissection. Relevant data included tumor-related variables, perioperative parameters, postoperative drainage status, postoperative subjective pain, and analgesic consumption amount were recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 80 years scheduled to receive neck dissection due to head and neck cancer

Exclusion Criteria:

* history of coagulation disorders
* prior radiation to the neck
* prior neck dissection
* declined to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shih-An Liu, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin WJ, Wang CC, Jiang RS, Huang YC, Ho HC, Liu SA. A prospective randomised trial of LigaSure Small Jaw(R) versus conventional neck dissection in head and neck cancer patients. Clin Otolaryngol. 2017 Apr;42(2):245-251. doi: 10.1111/coa.12702. Epub 2016 Jul 26. PMID 27390305

RESULTS

PARTICIPANT FLOW:
Groups:
- Ligusure-assisted Neck Dissection: The study group patients were treated using the LigaSure vessel sealing system (Small Jaw® with ForceTriad®; Covidien, Colorado, USA) for dissection and hemostasis throughout the whole procedures during neck dissection.
  Ligasure small jaw (Covidien, Colorado, USA): The Small Jaw® handpiece (Small Jaw® with ForceTriad®; Covidien, Colorado, USA) was not only used as a dissection forceps but also served as a ligation device.
- Conventional Neck Dissection: The control group patients were treated using conventional cold instrument dissection, monopolar electrocautery hemostasis, and suture ligation during neck dissection.
Period: Overall Study
Arm/Group | Ligusure-assisted Neck Dissection | Conventional Neck Dissection
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ligusure-assisted Neck Dissection | Conventional Neck Dissection | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (9.3) | 51.1 (8.1) | 52.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 16 | 18 | 34
Region of Enrollment [Number; unit: participants]
  Taiwan | 21 | 20 | 41
Primary tumor site [Number; unit: participants]
  Oral cavity | 12 | 12 | 24
  Oropharynx | 3 | 3 | 6
  Thyroid gland | 3 | 2 | 5
  Others | 3 | 3 | 6
Clinical N stage [Number; unit: participants] — Clinical N stage was in accordance with the guidelines of the American Joint Committee on Cancer (7th edition, 2009)
  Briefly, the clinical N stage was described at below.
  N0: No regional lymph node metastasis
  N1: Metastasis in a single ipsilateral lymph node, 3 cm or less in greatest dimension
  N2: Metastasis of regional lymph node(s), none more than 6 cm in greatest dimension
  Basically, a better survival is expected in N0 stage yet a worse survival is anticipated in N2 stage.
  participants
    N0 | 8 | 11 | 19
    N1 | 6 | 2 | 8
    N2 | 7 | 7 | 14
Levels of neck dissection [Number; unit: participants] — Level of cervical lymph node is based on the anatomical location
  Briefly, the level of cervical lymph node is described as below
  Level I: Submental and submandibular nodes
  Level II: Upper jugular nodes - Between posterior belly of digastric muscles superiorly and hyoid bone inferiorly
  Level III: Middle jugular nodes - between the hyoid bone and cricoid cartilage
  Level IV: Lower jugular nodes - between the cricoid cartilage and the clavicle
  Level V: Posterior cervical or spinal accessory nodes, posterior to the sternocleidomastoid muscle
  participants
    Level I, II, III | 12 | 14 | 26
    Level I, II, III, IV | 3 | 3 | 6
    Level II, III, IV | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Opreation Duration
Description: The duration from incision of cervial skin till the completion of lymph node dissection
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ligusure-assisted Neck Dissection | Conventional Neck Dissection
Number analyzed (Participants) | 21 | 20
minutes | 97.1 (22.5) | 116.3 (28.6)
Statistical Analysis 1: Comparison: Ligusure-assisted Neck Dissection vs Conventional Neck Dissection; Test type: Non-Inferiority or Equivalence — A previous study found that the mean operation time was 165 minutes for patients undergoing LigaSure vessel sealing system-assisted total laryngectomy plus neck dissection and 195 minutes for those receiving conventional hemostasis. With a difference in operative duration of 30 minutes between the two groups,9 the estimated sample size needed to demonstrate a two-sided significance level of 0.05 with 80% power should be at least 18 participants in each treatment arm; p = 0.022, t-test, 2 sided

2. Secondary Outcome: Intraoperative Blood Loss
Description: Intraoperative blood loss was estimated by the sum of the volume in the suction bottle and the increased weight of wet gauzes containing blood after neck dissection.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Ligusure-assisted Neck Dissection | Conventional Neck Dissection
Number analyzed (Participants) | 21 | 20
ml | 122 (63) | 144 (61)
Statistical Analysis 1: Comparison: Ligusure-assisted Neck Dissection vs Conventional Neck Dissection; Test type: Non-Inferiority or Equivalence — As above; p = 0.266, t-test, 2 sided

3. Secondary Outcome: Postoperative Drainage Amount
Description: The amount of drainage from closed system drainage tube
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Ligusure-assisted Neck Dissection | Conventional Neck Dissection
Number analyzed (Participants) | 21 | 20
ml | 107 (47) | 139 (58)
Statistical Analysis 1: Comparison: Ligusure-assisted Neck Dissection vs Conventional Neck Dissection; Test type: Non-Inferiority or Equivalence — as above; p = 0.060, t-test, 2 sided

4. Secondary Outcome: Postoperative Subjective Pain Status
Description: Visual analogue scale of subjective pain status after operation
Time Frame: 2 weeks
Population: Pain visual analogue scale (VAS) (no pain: 0, intolerable pain: 10)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ligusure Assisted Neck Dissection: The study group patients were treated using the LigaSure vessel sealing system (Small Jaw® with ForceTriad®; Covidien, Colorado, USA) for dissection and hemostasis throughout the whole procedures during neck dissection.
  Participants were asked to take a Voren enteric-microencapsulated (Diclofenac 50 mg/capsule) capsule 3 times a day for pain relief postoperatively. An additional capsule before sleep was allowed if persistent pain was told by the patient. When intolerable pain was complained in spite of oral analgesic, pethidine (meperidine 50 mg/ampule) injection was prescribed every 6 hours.
  Neck dissection: The Small Jaw® handpiece (Small Jaw® with ForceTriad®; Covidien, Colorado, USA) was not only used as a dissection forceps but also served as a ligation device.
- Conventional Neck Dissection: The control group patients were treated using conventional cold instrument dissection, monopolar electrocautery hemostasis, and suture ligation during neck dissection.
  Participants were asked to take a Voren enteric-microencapsulated (Diclofenac 50 mg/capsule) capsule 3 times a day for pain relief postoperatively. An additional capsule before sleep was allowed if persistent pain was told by the patient. When intolerable pain was complained in spite of oral analgesic, pethidine (meperidine 50 mg/ampule) injection was prescribed every 6 hours.
  Neck dissection: The Small Jaw® handpiece (Small Jaw® with ForceTriad®; Covidien, Colorado, USA) was not only used as a dissection forceps but also served as a ligation device.
Arm/Group | Ligusure Assisted Neck Dissection | Conventional Neck Dissection
Number analyzed (Participants) | 21 | 20
units on a scale
  Baseline | 0.6 (1.5) | 0.7 (1.2)
  6 hours after OP | 3.5 (2.5) | 3.4 (2.1)
  12 hours after OP | 2.5 (1.6) | 2.6 (1.7)
  1 day after OP | 2.5 (1.9) | 1.9 (1.7)
  3 days after OP | 2.3 (2.0) | 1.9 (1.7)
  7 days after OP | 1.2 (1.4) | 1.4 (2.2)
  14 days after OP | 0.7 (1.1) | 0.7 (1.3)

5. Secondary Outcome: Postoperative Oral Analgesic Consumption
Description: The amount of analgesic consumption via oral ingestion after operation
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: capsules
Arm/Group | Ligusure-assisted Neck Dissection | Conventional Neck Dissection
Number analyzed (Participants) | 21 | 20
capsules | 37.2 (15.6) | 40.9 (20.7)
Statistical Analysis 1: Comparison: Ligusure-assisted Neck Dissection vs Conventional Neck Dissection; Test type: Non-Inferiority or Equivalence — as above; p = 0.524, t-test, 2 sided

6. Secondary Outcome: Postoperative Injected Analgesic Amount
Description: The amount of injected form analgesic used (Meperidine 50 mg/ampule)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Ampule
Arm/Group | Ligusure-assisted Neck Dissection | Conventional Neck Dissection
Number analyzed (Participants) | 21 | 20
Ampule | 8.8 (11.3) | 17.7 (14.9)
Statistical Analysis 1: Comparison: Ligusure-assisted Neck Dissection vs Conventional Neck Dissection; Test type: Non-Inferiority or Equivalence — as above; p = 0.037, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 14 days after operation
Arm/Group | Ligusure-assisted Neck Dissection | Conventional Neck Dissection
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No